CLINICAL TRIAL: NCT00570245
Title: A Pilot, Single Center Prospective, With Parallel Groups, Controlled and Open to Evaluate the Efficacy of Nitric Oxide for Inhalation in Lung Donors and in the Prevention of Reperfusion Injury.
Brief Title: Safety and Efficacy Study of Nitric Oxide in Patients Going Through Lung Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VICER1
Record Dates: First submitted 2007-12-06; First posted 2007-12-10 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Lung Transplantation
Keywords: Lung transplantation
MeSH Terms: interventions — Nitric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (No Intervention): Neither donors or recipients will receive NO
- B (Active Comparator): Donor will not receive NO, recipient will receive up to 48 hours of NO
  Interventions: Drug: Nitric oxide
- C (Active Comparator): The donor will receive NO for 3 hours and the recipient will receive NO for up to 48 hours
  Interventions: Drug: Nitric oxide

INTERVENTIONS:
Drug: Nitric oxide — inhalation, 10 ppm, for up to 48 hours
  Arms: B
Drug: Nitric oxide — inhalation; 10ppm; 3 hours (donor) up to 48 hours (recipient)
  Arms: C

SUMMARY:
The purpose of this study is to assess the safety and efficacy of inhaled nitric oxide in prevention of lung graft dysfunction due to ischemia-reperfusion

DETAILED DESCRIPTION:
* Pilot, single-center, prospective, randomized, parallel-group, controlled, open-label trial.
* Sixty lung donors will be analyzed, making a comparative study between donors receiving NO for 3 hours prior to removal of the organ versus a control group to which NO will not be administered.
* A Swan-Ganz catheter will be placed to determine PVR, PAP, MV, and PCP; and blood gases will be done after arterial cannulation to determine FiO2/PaO2 hourly. Also, standard blood chemistry, hematology, coagulation parameters, and arterial blood gas.
* Prior to NO administration and before procurement, a BAL (bronchoalveolar lavage) will be done to determine the presence of leukocytes, predominantly neutrophils, IL-1, IL-6, IL-8, IL-10, TNF, and proteins as well as obtaining secretions for culture.
* The dosage of NO will be 10ppm, with NO2 and methemoglobinemia being monitored exhaustively.
* In the operating room and prior to lung removal, a new BAL will be done and the anti-inflammatory agents described above will be determined.
* Organ removal and the preservation fluid used will be standard, according to the established surgical protocol.
* Anesthesia: methylprednisolone 1 g will be administered before organ extraction; hemodynamic determinations of mAP, PAP, CVP, MV, and hourly urinary output and arterial blood gas.
* Hemodynamic and respiratory determinations will be made in the lung receptors: mAP, mPAP, PVR, MV, PCP, DO2, Qs/Qt, and CVP as well as gas determinations every 30 minutes, blood chemistry, hematology, and coagulation immediately after reperfusion. A BAL will also be done after anesthesia induction.
* Incidents during surgery will be recorded, especially the need for extracorporeal circulation as well as transfusion requirements and ischemia times.
* After surgery, another BAL will be done both 24 hours and 48 hours after return to the Recovery Unit. Hemodynamic and respiratory parameters will be monitored every 4 hours for the first 48 hours after surgery, as well as arterial blood gases.
* Blood chemistry will be done every 12 hours along with coagulation and hematology tests.
* Chest x-ray on admission and daily to determine the degree of the patient's edema over the first 48 hours.
* Drug administration: the NO will be administered in the respirator intake at a dose of 10ppm for 48 hours. A monitor will be used showing the gas dosage continuously, as well as NO2 and methemoglobinemia.
* The inflammatory agents (TNF, IL-1, IL-2, IL-6, IL-8, and IL-10) will be determined with the ELISA technique.

ELIGIBILITY:
Inclusion Criteria:

* Have a lung graft scheduled
* Males and females aged 18 to 65
* Signed informed consent approved by the IRB/EC

Exclusion Criteria:

* Uncontrolled bacterial infection
* Creatinine clearance <50 ml/min
* Severe extrapulmonary organic dysfunction
* Continuing smoking habit
* Neoplastic disease (2-5 years free of tumor, depending on type)
* Pregnancy or nursing
* Severe osteoporosis
* Active peptic ulcer
* Progressive neuromuscular disease
* Active limiting systemic disease. Complicated diabetes.
* Any contraindication based on the judgement of the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2005-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Edema and mPAP | 4 - 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Rosario Vicente, MD, Principal Investigator — Hospital General La Fe
Locations (1):
- Hospital General La Fe, Valencia, Spain

REFERENCES:
- [Background] Moreno I, Vicente R, Ramos F, Vicente JL, Barbera M. Determination of interleukin-6 in lung transplantation: association with primary graft dysfunction. Transplant Proc. 2007 Sep;39(7):2425-6. doi: 10.1016/j.transproceed.2007.07.056. PMID 17889209
- [Background] Moreno I, Mir A, Vicente R, Pajares A, Ramos F, Vicente JL, Barbera M. Analysis of interleukin-6 and interleukin-8 in lung transplantation: correlation with nitric oxide administration. Transplant Proc. 2008 Nov;40(9):3082-4. doi: 10.1016/j.transproceed.2008.08.124. PMID 19010201
- [Background] Moreno I, Vicente R, Mir A, Leon I, Ramos F, Vicente JL, Barbera M. Effects of inhaled nitric oxide on primary graft dysfunction in lung transplantation. Transplant Proc. 2009 Jul-Aug;41(6):2210-2. doi: 10.1016/j.transproceed.2009.05.019. PMID 19715875